CLINICAL TRIAL: NCT02475239
Title: Efficacy of Postural Restriction in Treating Benign Paroxysmal Positional Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Yuvatiya Plodpai, Doctor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 57-0082-13-1
Record Dates: First submitted 2015-06-10; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Benign Paroxysmal Positional Vertigo, Postural Restriction
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postural restriction (Experimental): The patients were instructed to avoid head movements, wear a soft collar during the daytime, wear a supporting pillow and sleep in the semi-upright position at a 45 degree head elevation from the horizontal plane during the nighttime for 48 hours.
  Interventions: Behavioral: Postural restriction
- Normal daily activity (Active Comparator): The patients did not follow any postural restrictions and were asked to live as normally as possible.
  Interventions: Behavioral: Normal daily activity

INTERVENTIONS:
Behavioral: Postural restriction — The patients were instructed to avoid head movements, wear a soft collar during the daytime, wear a supporting pillow and sleep in the semi-upright position at a 45 degree head elevation from the horizontal plane during the nighttime for 48 hours.
  Arms: Postural restriction
Behavioral: Normal daily activity — The patients did not follow any postural restrictions and were asked to live as normally as possible.
  Arms: Normal daily activity

SUMMARY:
The standard treatment of posterior semicircular canal benign paroxysmal positional vertigo is the canalith repositioning procedure or the Epley maneuver. Based on the present literature, there is controversy on the efficacy of post-maneuver postural restrictions.The aim of this study was to conduct a randomized controlled trial to compare the treatment efficacy of post-maneuver postural restriction with CRP alone in patients with posterior semicircular canal benign paroxysmal positional vertigo.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo is the most common cause of vertigo. Based on the present literature, there is controversy on the efficacy of post-maneuver postural restrictions.Some study designs were not randomized controlled trials. The present study offers an alternative way of postural restriction to maintain postural restriction as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral posterior semicircular canal benign paroxysmal positional vertigo and
* A negative neurologic examination

Exclusion Criteria:

* Secondary benign paroxysmal positional vertigo caused by trauma head injury, inner ear surgery, viral labyrinthitis or Meniere's disease
* Patients with central vertigo, cervical spine, neurologic, otologic, psychiatric diseases
* Patients who used medications that affected the neurologic and otologic systems for less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The Dix-Hallpike test | 2 weeks
  The Dix-Hallpike test results

SECONDARY OUTCOMES:
Resolution time | 24 weeks
  Time interval until the patient report recurrent vertigo confirmed by positive Dix-Hallpike
Medication needed | 24 weeks
  Need of medication to treat vertigo (in this study, betahistine)
the Dizziness Handicap Inventory (DHI) | 24 weeks
Recurrent rate | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuvatiya Plodpai, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Yuvatiya Plodpoai, Hat Yai, Changwat Songkhla, Thailand